Pilot Study on a Health Promotion Intervention for Ultra-Orthodox Mothers of Children With ADHD

NCT06703242

Date: January 30, 2024

# **Explanation and Consent Form for Participation in Research Study Titled:**

# Pilot Study on a Health Promotion Intervention for Ultra-Orthodox Mothers of Children With ADHD

## **Background and Purpose of the Research:**

Mothers of children with ADHD in the Ultra-Orthodox community often experience stress and are at risk of related challenges. Therefore, a group intervention program tailored to the community's needs has been developed to promote the health of these mothers.

This study, conducted by the Hebrew University's School of Occupational Therapy, aims to evaluate the effectiveness of this group intervention for Ultra-Orthodox mothers of children with ADHD.

The results of this study may contribute to improving the health and well-being of these mothers.

#### **Eligibility Criteria:**

#### 1. Mothers:

 Mothers of a child aged 6–12 diagnosed with ADHD, belonging to the Ultra-Orthodox community, and with no other significant family health conditions (apart from ADHD).

#### 2. Educators:

- Educators with experience teaching at least five children diagnosed with ADHD in elementary schools within the Ultra-Orthodox community.
- The educator does not represent any specific organization or institution but acts as an independent expert in the field of education for children with ADHD.

## **What Participation Involves:**

#### **For Mothers:**

- 1. Participation in a six-session group program (90 minutes per session) via Zoom, held weekly with 6–8 mothers per group.
- 2. Completion of questionnaires before and after the program (approximately 30 minutes each).
- 3. Participation in a 90-minute focus group to provide feedback after the program via Zoom.

#### For Educators:

- 1. Participation in a single group session (90 minutes) during the program via Zoom.
- 2. Participation in a 90-minute interview to provide feedback after the program via Zoom.

#### **Important Notes:**

- Sessions, focus groups, and interviews will be conducted by researchers Jennifer Budman and Prof. Adina Maeir.
- Sessions will be recorded for transcription purposes. The recordings will be stored securely and deleted after transcription. Participants are advised to participate in a private, quiet location to ensure confidentiality.

#### **Participant Declaration:**

#### 1. Potential Benefits:

This study will assist in evaluating the feasibility of a health promotion intervention for mothers of children with ADHD.

#### 2. Institutional Support:

The study is conducted under the School of Occupational Therapy at the Hebrew University of Jerusalem, within the Neurocognitive Rehabilitation Lab led by Prof. Adina Maeir. For questions, participants may contact Jennifer Budman at 050-3422600 or Jennifer.budman@mail.huji.ac.il, or Prof. Adina Maeir at 054-6205081 or adina.maeir@mail.huji.ac.il.

## 3. Voluntary Participation:

I am free to choose not to participate and can withdraw from the study at any time without affecting my rights.

#### 4. Right to Refuse Questions:

I have the right to refrain from answering any questions I do not wish to answer.

#### 5. Consultation:

I have the right to consult with others (e.g., family members) before deciding to participate in this study.

# 6. Confidentiality in Group Settings:

While participants will be asked to respect the privacy of others during group sessions, full confidentiality cannot be guaranteed due to the group setting.

#### 7. Recording of Focus Groups:

I understand that focus groups will be recorded. The recordings will be saved as password-protected files on the researcher's private computer (not cloud storage) for up to one month for transcription purposes, without identifiable details, and will then be permanently deleted.

## 8. Anonymity and Data Use:

Recordings and transcripts will remain confidential and accessible only to the researchers, Jennifer Budman and Prof. Adina Maeir. The data collected will not include identifying information and will be coded for anonymity.

# 9. Purpose of Data Collection:

I understand that the data collected is solely for research purposes.

#### 10. Risks and Discomfort:

Participation in this study poses no physical risks. However, participants may experience some discomfort during questionnaires or sessions, either due to the time required or the nature of certain reflective questions.

#### 11. Consent to Participate:

By signing this form, I consent to participate in the study, including completing questionnaires, attending program sessions, providing feedback in focus groups (for mothers), or participating in feedback interviews (for educators). I also consent to the recording of sessions for data collection purposes.

| Date: | Signature: |
|-------|------------|
|-------|------------|